CLINICAL TRIAL: NCT01951768
Title: A Randomized, Controlled Study to Investigate the Efficacy and Safety of a Topical Gentamicin-Collagen Sponge in Combination With Systemic Antibiotic Therapy in Diabetic Patients With a Moderate or Severe Foot Ulcer Infection
Brief Title: Efficacy and Safety of Garamycin® Sponge in Diabetic Patients With a Moderate or Severe Foot Ulcer Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Ilker Uckay, Consultant Service of Infectious Diseases, Consultant for Septic Orthopaedics, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUG protocol
Record Dates: First submitted 2013-09-18; First posted 2013-09-27 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Garamycin Sponge (Gentamicin-Collagen Sponge) (Experimental): Garamycin Sponge (Gentamicin-Collagen sponge) applied daily plus systemic antibiotic and standard ulcer care
  Interventions: Drug: Garamycin Sponge (Gentamicin-Collagen sponge)
- Systemic Antibiotic (Active Comparator): Systemic antibiotic therapy and standard ulcer care
  Interventions: Drug: Systemic Antibiotic

INTERVENTIONS:
Drug: Garamycin Sponge (Gentamicin-Collagen sponge) — Gentamicin Collagen Sponge: 5 × 5 cm in size containing Type I bovine collagen and 50 mg of gentamicin sulfate (equivalent to 32.5 mg of gentamicin base)
  Other Names: Sponge arm
  Arms: Garamycin Sponge (Gentamicin-Collagen Sponge)
Drug: Systemic Antibiotic — Antibiotics options per protocol:
  Levofloxacin PO 750 mg q.24h or 500 mg q.12h Levofloxacin IV 750 mg q.24h or 500 mg q.12h Amoxicillin/clavulanate PO 500/125 mg q.12h. or q.8h Amoxicillin/clavulanate IV 1000/200 mg q.12h or q.8h Clindamycin PO 300 mg or 450 mg q.6h Clindamycin IV 600 mg q.8h or q.6h Linezolid PO 600 mg q.12h Linezolid IV 600 mg q.12h Metronidazole PO 400 mg or 500 mg q.8h or 500 mg q.6h Metronidazole IV 500 mg q.8h or q.6h Aztreonam IV 1 g or 2 g q.12h or q.8h Piperacillin/tazobactam IV 3000/375 mg q.6h or 4000/500 mg q.8h
  Other Names: Control arm
  Arms: Systemic Antibiotic

SUMMARY:
The purpose of this study is to determine whether Garamycin Sponge (Gentamicin-Collagen sponge) in combination with antibiotics is safe and effective in treating moderate and severe diabetic foot infections.

DETAILED DESCRIPTION:
Infected skin ulcers with diabetes can be very debilitating because they are difficult to heal. Diabetic ulcers are responsible for frequent health care visits, and are a major predictor of amputation. Diabetic ulcers can be caused by a patient's inability to sense pain or warmth as well as peripheral vascular disease, which causes diminished blood flow to the foot. Early aggressive treatment is necessary to treat infection and ultimately prevent the need for amputation.

Gentamicin is an antibiotic that is effective in treating certain kinds of infection. Collagen is a protein that is found in all mammals. The gentamicin sponge being used in this study is commercially available in Switzerland as Garamycin® Sponge. The Garamycin Sponge is a thin flat sponge made out of collagen that comes from bovine tendons and containing gentamicin. When applied to an open ulcer, the collagen breaks down and the gentamicin is released into the ulcer, but very little is absorbed into the blood stream. The high levels of gentamicin in the open infected ulcer may help treat the infection.

All subjects will be given the necessary supplies and taught how to take care their foot ulcer. All subjects will also receive oral an antibiotic. Additionally, subjects who are randomly assigned to receive the gentamicin-collagen sponge will place a gentamicin-collagen sponge on their ulcer during daily wound care.

ELIGIBILITY:
Inclusion Criteria:

* Is aged ≥ 18.
* Has diabetes mellitus, according to the American Diabetes Association (ADA) criteria.
* Has an open foot wound with visible inflammation, namely at least 1 skin ulcer located on or below the malleolus that presents with the following clinical manifestations of a moderate or severe infection based on the Infectious Disease Society of America (IDSA).
* Has received appropriate surgical intervention to remove all necrotic and infected bone if diagnosed with osteomyelitis
* Meets certain minimal laboratory criteria.

Exclusion Criteria:

* Has an ulcer infection which, based upon the patient's known history of hypersensitivity cannot be appropriately treated with at least one of the empiric systemic antibiotic regimens per protocol.
* Has received > 48 hours of potentially effective antibiotic therapy and the wounds are clinically improving. If a patient has received an antibiotic within 72 hours, but is not improving or deep-tissue culture results indicate that the infecting pathogen is not susceptible to that antibiotic, the patient may be enrolled.
* Requires or is likely to require treatment with any concomitant topical product or wound therapy during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Background] Uckay I, Kressmann B, Malacarne S, Toumanova A, Jaafar J, Lew D, Lipsky BA. A randomized, controlled study to investigate the efficacy and safety of a topical gentamicin-collagen sponge in combination with systemic antibiotic therapy in diabetic patients with a moderate or severe foot ulcer infection. BMC Infect Dis. 2018 Aug 2;18(1):361. doi: 10.1186/s12879-018-3253-z. PMID 30068306
- [Background] Uckay I, Kressmann B, Di Tommaso S, Portela M, Alwan H, Vuagnat H, Maitre S, Paoli C, Lipsky BA. A randomized controlled trial of the safety and efficacy of a topical gentamicin-collagen sponge in diabetic patients with a mild foot ulcer infection. SAGE Open Med. 2018 May 13;6:2050312118773950. doi: 10.1177/2050312118773950. eCollection 2018. PMID 29785265

RESULTS

PARTICIPANT FLOW:
Groups:
- Systemic Antibiotic: Systemic antibiotic therapy and standard ulcer care
  Systemic Antibiotic: Antibiotics options per protocol:
  Levofloxacin PO 750 mg q.24h or 500 mg q.12h Levofloxacin IV 750 mg q.24h or 500 mg q.12h Amoxicillin/clavulanate PO 500/125 mg q.12h. or q.8h Amoxicillin/clavulanate IV 1000/200 mg q.12h or q.8h Clindamycin PO 300 mg or 450 mg q.6h Clindamycin IV 600 mg q.8h or q.6h Linezolid PO 600 mg q.12h Linezolid IV 600 mg q.12h Metronidazole PO 400 mg or 500 mg q.8h or 500 mg q.6h Metronidazole IV 500 mg q.8h or q.6h Aztreonam IV 1 g or 2 g q.12h or q.8h Piperacillin/tazobactam IV 3000/375 mg q.6h or 4000/500 mg q.8h
Period: Overall Study
Arm/Group | Garamycin Sponge (Gentamicin-Collagen Sponge) | Systemic Antibiotic
Started | 43 | 45
Completed | 43 (43 patients) | 45 (45 patients)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There are no protocol violations leading to a change in the number of assigned patients in either study arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Garamycin Sponge (Gentamicin-Collagen Sponge) | Systemic Antibiotic | Total
Number analyzed (Participants) | 43 | 45 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 22 | 43
  >=65 years | 22 | 23 | 45
Age, Continuous [Median (Standard Deviation); unit: years] | 71 (8) | 72 (8) | 71 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 27 | 28 | 55
Region of Enrollment [Number; unit: participants]
  Switzerland | 43 | 45 | 88

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure
Description: Clinical Cure defined as the absence of any clinical, radiological or laboratory evidence of infection
Time Frame: Approximately day 38
Measure: Number; unit: participants
Arm/Group | Garamycin Sponge (Gentamicin-Collagen Sponge) | Systemic Antibiotic
Number analyzed (Participants) | 43 | 45
participants | 38 | 39

2. Secondary Outcome: Clinical Response
Description: Clinical significant improvement is defined as significant improvement of infection but not complete cure (e.g., residual uninfected skin lesions).
Time Frame: up to 38 days
Measure: Number; unit: participants
Arm/Group | Garamycin Sponge (Gentamicin-Collagen Sponge) | Systemic Antibiotic
Number analyzed (Participants) | 43 | 45
participants | 7 | 13

3. Secondary Outcome: Pathogen Eradication
Description: Microbiological eradication of former infection
Time Frame: up to 38 days
Measure: Number; unit: participants
Arm/Group | Garamycin Sponge (Gentamicin-Collagen Sponge) | Systemic Antibiotic
Number analyzed (Participants) | 43 | 45
participants | 26 | 20

ADVERSE EVENTS:
Arm/Group | Garamycin Sponge (Gentamicin-Collagen Sponge) | Systemic Antibiotic
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45
Other Adverse Events (participants affected / at risk) | 0/43 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes